CLINICAL TRIAL: NCT06977893
Title: Neoadjuvant Chemotherapy in Combination With Toripalimab for HR+/HER2- Breast Cancer : a Randomized, Open-label, Parallel-controlled, Multi-center Phase III Study (NEOTORCH-BREAST04)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250026C
Record Dates: First submitted 2025-05-12; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: HR+/HER2- Breast Cancer
Keywords: Breast cancer; Toripalimab; Adjuvant Chemotherapy; Immunotherapy; HR-positive HER2-negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Neoadjuvant Chemotherapy in Combination with Toripalimab (Experimental): Drug: Neoadjuvant Chemotherapy in Combination with Toripalimab Description: Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks. During neoadjuvant chemotherapy and postoperative adjuvant therapy, use of Toripalimab: intravenous infusion of 240 mg, once every 3 weeks, combined with preoperative neoadjuvant and postoperative adjuvant therapy for a total of 1 year.
  Interventions: Drug: Neoadjuvant Chemotherapy in Combination with Toripalimab
- Control Group: Neoadjuvant Chemotherapy (Sham Comparator): Drug: Neoadjuvant Chemotherapy Description: Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks.
  Interventions: Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy in Combination with Toripalimab — Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks. During neoadjuvant chemotherapy and postoperative adjuvant therapy, use of Toripalimab: intravenous infusion of 240 mg, once every 3 weeks, combined with preoperative neoadjuvant and postoperative adjuvant therapy for a total of 1 year.
  Arms: Experimental Group: Neoadjuvant Chemotherapy in Combination with Toripalimab
Drug: Neoadjuvant Chemotherapy — Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks.
  Arms: Control Group: Neoadjuvant Chemotherapy

SUMMARY:
Our center plans to conduct a randomized, open-label, parallel-controlled, multi-center phase III study to evaluate the efficacy and safety of neoadjuvant chemotherapy combined with Toripalimab for HR+/HER2- breast cancer. The aim is to further explore the treatment strategy of chemotherapy with immunotherapy for patients with HR+/HER2- breast cancer, provide more treatment options for breast cancer patients, and offer a potential theoretical basis for the precision treatment of breast cancer.The primary study objective is to evaluate the pathologic complete response（PCR）and RCB0-1 ratio of neodjuvant treatment of HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years old;
2. ECOG score is 0-1 points;
3. breast cancer meets the following standards: Histologically confirmed invasive breast cancer with tumor diameter>1cm (T1c-3; N0-3; M0). All patients were pathohistologically confirmed as HR+/HER2- breast cancer. According to the breast cancer diagnosis and treatment guidelines and specifications of the Chinese Anti Cancer Association (2021 version), Luminal B is divided into Luminal B (HER2 negative) and Luminal B (HER2 positive). Luminal B (HER2 negative) is ER/PR positive, HER2 negative and Ki-67 proliferation index is high or PR low expression. Luminal type B (HER2 positive) is ER/PR positive, HER2 positive (protein overexpression or gene amplification), and Ki-67 in any state. Therefore, HR+/HER2- breast cancer is a Luminal type breast cancer patient excluding HER2+.

   Pathological examination of PD-L1 expression:

   The Combined Positive Score (CPS) refers to the percentage of PD-L1 positive cells (including tumor cells, lymphocytes, macrophages) in all tumor cells. Our center detected the PD-L1 antibody site as 22C3.
4. The functional level of major organs must meet the following requirements (no blood transfusion within 2 weeks before screening, no use of...)

Using leukocyte and platelet boosting drugs:

1. Blood routine: Absolute neutrophil count (ANC) greater than 1.5 × 109/L; platelet count (PLT) greater than 75 × 109/L; Hemoglobin (Hb) is greater than 90g/L; Lymphocyte count ≥ 1.5 × 109/L
2. Blood biochemistry: Total bilirubin (TBIL) is less than 1.5 × ULN; Alanine aminotransferase ALT and aspartate levels are less than 1.5 × ULN; Alkaline phosphatase is less than 2.5 × ULN; Urea nitrogen/ Urea (BUN/UREA) and creatinine (Cr) are less than 1.5 × ULN.
3. Cardiac ultrasound: Left ventricular ejection fraction (LVEF) greater than 55%.
4. 12 lead electrocardiogram: The Fridericia corrected QT interval (QTcF) is less than 470 milliseconds 5. For female patients who have not yet reached menopause or undergone surgical sterilization: during the treatment period and in the study treatment, the final use effective contraceptive methods for at least 6 months after a single administration.

6. Voluntarily join this study, sign an informed consent form, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Stage IV breast cancer.
2. Inflammatory breast cancer.
3. Previously received anti-tumor treatment or radiation therapy for any malignant tumor, excluding those that have been cured Malignant tumors such as cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma.
4. Simultaneously undergoing anti-tumor treatment in other clinical trials, including but not limited to chemotherapy and endocrine therapy. Treatment, biological therapy, bone improvement drug therapy, or immune checkpoint inhibitor therapy, etc.
5. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before the first administration of the study drug, or the patient has not fully recovered from such surgical procedures.
6. Serious heart disease or discomfort, including but not limited to the following diseases:

1) Diagnosed history of heart failure or systolic dysfunction (LVEF less than 50%).

2) High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate greater than 100bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block (i.e. Mobitz II second or third degree atrioventricular block).

3) Angina requiring medication for treatment. 4) Heart valve disease with clinical significance. 5) ECG shows transmural myocardial infarction. 6) Poor control of hypertension (systolic blood pressure greater than 180mmHg and/or diastolic blood pressure greater than 180mmHg after drug treatment) 100mmHg). 7. Uncontrolled active infections that require treatment; History of immunodeficiency, including HIV testing positive Sexual, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

8. Patients with chronic active hepatitis B or active hepatitis C (excluding hepatitis B virus carriers, stable hepatitis B after drug treatment [HBV-DNA test negative or<50IU/ml] and cured hepatitis C patients [HCV RNA test negative]).

9. Have received immunotherapy and experienced adverse immune events such as immune related pneumonia and myocarditis, which have been determined by researchers to potentially affect the safety of the experimental medication.

10. Individuals with a known history of allergies to the components of this medication regimen.

11. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or reproductive age patients who are unwilling to take effective contraceptive measures during the entire trial period and within 6 months after the last study medication.

12. Suffering from serious accompanying diseases or other comorbidities that may interfere with the planned treatment, or any other circumstances that the researcher deems unsuitable for the patient to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-03-23 (Estimated); Study Completion 2030-03-23 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response（PCR） | 2 years
  The primary study objective is to evaluate the pathologic complete response（PCR） of the control group and experimental group.
RCB 0-1 Ratio | 2 years

SECONDARY OUTCOMES:
Event Free Survival（EFS) | 5 years
  Event Free Survival (EFS) refers to the time from the start of randomization (the start of treatment in a single-arm trial) to the first occurrence of any of the following events: disease progression that makes surgical treatment impossible, local or distant recurrence, death due to any cause, etc. It can be used to evaluate the effectiveness of the drug.
Objective Response Rate (ORR) | 5 years
  Objective Response Rate (ORR) is a key indicator used in medical research, especially in oncology, to evaluate the effectiveness of a treatment. It refers to the proportion of patients whose tumor volume shrinks to a certain extent and remains in that state for a specific period of time after receiving a particular treatment.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Jinhua Municipal Central Hospital, Jinhua
  - Nanchang People's Hospital, Nanchang
  - Nantong First People's Hospital, Nantong
  - Zhongshan Hospitall, Fudan University, Shanghai
  - Xinjiang Medical University Affiliated Cancer Hospital, Ürümqi
  - Shaanxi Provincial Cancer Hospital, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou